CLINICAL TRIAL: NCT06462417
Title: Study on the Efficacy and Safety of Oral Administration of Arbidol in the Treatment of Allergic Rhinitis Patients
Brief Title: Efficacy and Safety of Arbidol in the Treatment of Allergic Rhinitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zheng Liu (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Zheng Liu, Professor of Otolaryngology-Head & Neck Surgery Vice Director Department of ENT Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Arbidol-01
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — umifenovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arbidol (Experimental): Arbidol Hydrochloride Tablets
  Interventions: Drug: Arbidol

INTERVENTIONS:
Drug: Arbidol — Arbidol Hydrochloride Tablets 0.2g/d for 2 weeks
  Other Names: Arbidol Hydrochloride

SUMMARY:
The most important treatment for AR is topical nasal medications (including nasal corticosteroids, nasal antihistamines, nasal decongestants, and nasal saline irrigation etc.), which are still limited. Arbidol may inhibit molecular targets involved in the pathogenesis of AR. This study intends to explore the effect of Arbidol in the treatment of allergic rhinitis and evaluate its efficacy and safety.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is a non-infectious inflammatory disease of the nasal mucosa mediated by Immunoglobulin E after exposure to allergens. AR has become a major chronic inflammatory disease of the respiratory tract, which has a serious impact on the quality of life of patients and social economy. The most important treatment for AR is topical nasal medications (including nasal corticosteroids, nasal antihistamines, nasal decongestants, and nasal saline irrigation etc.). However, even if patients are treated completely according to the standard diagnosis and treatment strategy, a considerable number of patients still do not achieve satisfactory treatment results. Arbidol is a medicine for the prevention and treatment of influenza. Based on our previous laboratory data, Arbidol may inhibit molecular targets involved in the pathogenesis of AR. In order to make the treatment of AR more effective, timely and convenient, this study intends to explore the effect of Arbidol in the treatment of allergic rhinitis and evaluate its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with allergic rhinitis (in line with the diagnostic criteria of the "Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (2015, Tianjin)" formulated by the Rhinology Group of the Otolaryngology-Head and Neck Surgery Branch of the Chinese Medical Association).
* 2. At least 2 nasal symptoms are moderate or above (referring to sneezing, runny nose, nasal itching, nasal congestion with at least 2 symptoms ≥2 points).
* 3. Female subjects are not pregnant or lactating and have no pregnancy and lactation plans during the trial medication period.
* 4. The subject has not participated in other clinical trials in the previous three months and agrees not to participate in other clinical trials before reaching the endpoint of this trial.
* 5. The subject/legally authorized representative understands the purpose and procedures of the trial and voluntarily signs the informed consent form, voluntarily participates in the study and complies with the study regulations, understands and complies with the medication dosage and follow-up plan, and correctly records the scale score, the number of medications, concomitant medication and adverse event records.

Exclusion Criteria:

* 1. Who are allergic to Arbidol.
* 2. Patients with abnormal liver and kidney function (ALT and AST exceed the maximum limit of normal value by 1.5 times, and Cr exceeds the upper limit of normal value).
* 3. Patients with abnormal ECG parameters and clinically significant (PR>220ms, QRS>120ms, QTc>450ms) and bradycardia.
* 4. Patients with severe asthma or acute asthma exacerbations.
* 5. Patients with structural heart disease, severe hypertension (blood pressure greater than 180/110mmHg), diabetes, hyperthyroidism, malignant tumors, immunocompromise, and mental illness. Patients with structural heart disease, severe hypertension (blood pressure greater than 180/110mmHg), diabetes, hyperthyroidism, malignant tumors, immunocompromise, and mental illness.
* 6. Patients with nasal polyps, severe deviated nasal septum, sinusitis, and hypertrophic rhinitis.
* 7. Who have participated in other clinical studies within 3 months.
* 8. Women are pregnant or lactating, in childbearing age with positive blood pregnancy test, or have pregnancy and lactation plans during the trial medication.
* 9. Drug abuse and alcoholism.
* 10. Who have received allergen-specific immunotherapy within 3 years.
* 11. Positive infectious disease screening (hepatitis B surface antigen, hepatitis C antibody, AIDS antibody and treponema pallidum antibody).
* 12. Who should not be included if there are other reasons in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The protein level of molecular biomarkers in nasal epithelial cells | 14 days
  The level of molecular biomarkers in nasal epithelial cells at baseline (day 0, prior to treatment), day 14 will be measured by western blotting.
The mRNA level of inflammation molecular biomarkers in nasal epithelial cells | 14 days
  The relative mRNA level of inflammatory cytokines (including IL-4, IL-13, CCL11, CCL24, CCL26 etc.) in nasal epithelial cells at baseline (day 0, prior to treatment), day 14 will be measured by Real-time PCR.
The level of inflammation molecular biomarkers in nasal lavage fluid | 14 days
  Investigate the change of inflammation molecular biomarkers using sample of nasal lavage fluid. Biomarkers including IL-4, IL-13, CCL11, CCL24, CCL26 and IgE etc. in nasal lavage fluid at day 7 day 14 were detected to compare the changes of molecular indices relative to baseline at day 0.

SECONDARY OUTCOMES:
Changes from baseline in daily total nasal symptom score (TNSS) during 2 weeks of treatment. | 14 days
  The TNSS for allergic rhinitis was used to evaluate the rhinitis-related symptoms and quantity of life scores. Changes from baseline in daily total nasal symptom score (TNSS) during 2 weeks of treatment. The Total Nasal Symptom Score (TNSS) is the sum of four symptom scores, rhinorrhea, nasal congestion, nasal itching, and sneezing, where each symptom is scored on a scale of 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Liu, Doctor, Study Chair — Tongji Hospital
Locations (2):
- China (2):
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Department of ENT, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei